CLINICAL TRIAL: NCT04855630
Title: Combating Alzheimer's Through Sleep and Exercise (CASE)
Brief Title: Combating Alzheimer's Through Sleep and Exercise
Acronym: CASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Shipley Foundation (Unknown); Dreem (Industry)
Responsible Party: Principal Investigator, Azizi Seixas, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20220931; 20-01023 (Other: NYU)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sleep Only Group (Experimental): Participants in this group will wear the DREEM 2 headband for 12 weeks.
  Interventions: Device: DREEM 2 Headband
- Exercise Only Group (Active Comparator): Participants in this group will workout twice a week for 12 weeks.
  Interventions: Other: Exercise Routine
- Exercise and Sleep Group (Active Comparator): Participants in this group will take part in a guided exercise program in additional to wearing the DREEM 2 headband for 12 weeks.
  Interventions: Device: DREEM 2 Headband; Other: Exercise Routine

INTERVENTIONS:
Device: DREEM 2 Headband — Participants will wear the DREEM 2 headband for 3 months for a minimum of 4 out of 7 nights per week and will participate in its digital therapeutic Cognitive Behavioral Therapy - Insomnia (CBT-I) intervention (entails brain stimulation to improve slow wave sleep and sleep hygiene counseling tips to improve sleep behaviors).
  Arms: Exercise and Sleep Group; Sleep Only Group
Other: Exercise Routine — Participants will partake in a guided exercise routine. Each routine consists of 30-minute mild circuit training session twice per week for 3 months.
  Arms: Exercise Only Group; Exercise and Sleep Group

SUMMARY:
The purpose of this research is to see how sleep and exercise affects dementia risk over time.

ELIGIBILITY:
Inclusion Criteria:

1. Able to perform mild exercise
2. Able to wear DREEM 2 Headband
3. Able to wear a Fitbit wrist watch
4. Able to perform the Everlywell biomarker procedure
5. Able to Understand and Speak English
6. Able to operate a digital device like mobile phone, iPad, or computer
7. Self-reported history of problems with cognitive impairment: memory, concentration, and processing information
8. Only participants cognitively able and willing to provide consent will be included.

Exclusion Criteria:

1. Prohibited from or unable to perform mild exercise
2. Unable to wear wrist watch or headband devices, or unable to supply pinprick blood sample for any reason
3. Unable to speak or understand English
4. Unable to use mobile device/smartphone technology
5. Unable or unwilling to consent for any reason.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Total Cholesterol Levels | Up to Week 12
  Measured from blood sample
High-Density Lipoprotein (HDL) Levels | Up to Week 12
  Measured from blood sample
Low-Density Lipoprotein (LDL) Levels | Up to Week 12
  Measured from blood sample
Triglycerides Levels | Up to Week 12
  Measured from blood sample
High-sensitivity C-reactive protein (hs-CRP) Levels | Up to Week 12
  Measured from blood sample
HbA1c Levels | Up to Week 12
  Measured from blood sample
Heart Rate | Up to Week 12
  Measured from Fitbit
Blood Pressure | Up to Week 12
  Measured from Fitbit
Total Sleep Duration | Up to Week 12
  Measured from DREEM 2
Slow Wave Sleep Duration | Up to Week 12
  Measured from DREEM 2
Cortisol Levels | Up to Week 12
  Measured from Urine Sample
Cortisone Levels | Up to Week 12
  Measured from Urine Sample
Melatonin Levels | Up to Week 12
  Measured from Urine Sample
Creatinine Levels | Up to Week 12
  Measured from Urine Sample

CONTACTS AND LOCATIONS:
Overall Officials: Azizi A Seixas, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospitals, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No